CLINICAL TRIAL: NCT01566565
Title: The Safety Evaluation of Theophylline and Bambuterol When Administered Orally Alone and in Combination to Healthy Volunteers
Brief Title: The Safety Evaluation of Drug Combinations Against High Altitude Pulmonary Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norwegian Armed Forces Medical Service (Other Government)
Collaborators: Duke University (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trond-Eirik Strand, Assistant Director General, Norwegian Armed Forces Medical Service
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1-Strand
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: High Altitude Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary edema of mountaineers | interventions — Theophylline; bambuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theophylline (Active Comparator)
  Interventions: Drug: Theophylline and Bambuterol
- Bambuterol (Active Comparator)
  Interventions: Drug: Theophylline and Bambuterol

INTERVENTIONS:
Drug: Theophylline and Bambuterol — Treatment 3: Theophylline, 300 mg plus Bambuterol, 20 mg

SUMMARY:
This is a Phase I, three period, two sequence, open-label, randomized, crossover study, with the primary objective of testing the safety and tolerability of combined oral doses of theophylline and bambuterol in healthy human subjects. The secondary objective is to assess the pharmacokinetic profiles of theophylline and bambuterol when administered alone or in combination. It is hypothesized that the combination of these drugs is generally safe, and that no drug interaction can be observed.

DETAILED DESCRIPTION:
This is a Phase I, three period, two sequence, single-center, open-label, randomized, crossover study design. Periods I and II consist of the oral administration of either a single dose of theophylline or bambuterol alone, followed by a 7 day wash out interval. Subsequently, Period III consists of the simultaneous administration of both drugs. All subjects are to be confined to the Oslo University Hospital Research Unit throughout all treatment periods [Study Day 1, 7 and 14]. A sufficient number of healthy adult subjects will be consented in order to enroll 20 and complete 16 subjects who complete all three periods. Replacement of subjects is permitted, if necessary.

Qualified subjects will be randomized into one of two sequences consisting of three Periods as indicated below:

-------------Period 1-----Period 2-----Period 3

Sequence A: Treatment 1 Treatment 2 Treatment 3

Sequence B: Treatment 2 Treatment 1 Treatment 3

TREATMENTS:

Treatment 1: Theophylline 300 mg.

Treatment 2: Bambuterol 20 mg.

Treatment 3: Theophylline 300 mg plus Bambuterol 20 mg.

After completion of each treatment period, the subjects will proceed to the next period provided no Stopping Rules criteria have been met

ELIGIBILITY:
Inclusion criteria:

1. Subjects must give written informed consent to participation in the study prior to screening. Consent will be documented by the subject's dated signature
2. Subjects must be healthy non-smoking adult male and female volunteers between the ages of 18 and 40 years, with a BMI of 18-30 kg/m2 and weighing at least 68 kg. Subjects health status will be determined by the medical history, physical examination, vital signs, electrocardiogram, blood chemistry, hematology, and urinalysis performed at screening.
3. Subjects must be willing to fast a minimum of 8 hours prior to screening.
4. Subjects must be willing to abstain from alcohol and xanthine-containing food and beverages (in example coffee, tea, and colas) from 48 hours before the time of admission to the clinical research inpatient unit and until last PK sample of drug given on day 1, 7 and 14 is drawn after 24 hours.
5. Subjects must be willing to remain in the clinical research unit continuously for the inpatient portion of the study from admission to discharge.
6. Women who are of non-childbearing potential, must be:

   1. Surgically sterile (removal of both ovaries and/ or uterus at least 12 months prior to dosing)
   2. Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing on Day -1, with an FSH level at screening of ≥ 40 mIU/mL.
7. Women of child-bearing potential must have a negative serum pregnancy test within 48 hours of receiving study drug and must agree to avoid pregnancy during study and for one month after the last dose of study drug.
8. Female subjects of child-bearing potential must agree to avoid pregnancy during study and for three months after the last dose of study drug.
9. Subjects must agree not to donate blood, plasma, platelets, or any other blood components during the study and for 4 weeks after the last dose.
10. Male subjects must agree not to donate sperm during the study and for 12 weeks after the last dose.

Exclusion criteria

Individuals meeting ANY ONE of the following criteria will be excluded from the study:

1. Subjects with laboratory results outside the normal range, if considered clinically significant by the Investigator. In addition, subjects must have a normal hematocrit and hemoglobin concentration and be ≥ 36% and ≥ 12.0 g/dL, respectively and plasma potassium concentration of at least 3.9 mmol/l.
2. A mental capacity that is limited to the extent that the subject cannot provide legal consent or understand information regarding the side effects of the study drug.
3. Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years.
4. Unwillingness or lack of ability to comply with the protocol, or to reside in the inpatient unit during the required time period, or to cooperate fully with the Principle Investigator and site personnel.
5. Use of any of the following:

   1. Any concomitant medication including oral contraceptive hormones. Subjects who have received any prescribed or non-prescribed (over-the-counter [OTC]) systemic medication, topical medications, or herbal supplements within 14 days from Day 1. St. John's Wort (hypericin) must not have been taken for at least 30 days prior to Period 1, Day 1.
   2. Any drugs, foods or substances known to be strong inhibitors or strong inducers of CYP enzymes (also known as cytochrome P450 enzymes); especially CYP 1A2, or Pgp within 30 days prior to Period 1, Day 1.
6. Clinically significant ECG abnormality in the opinion of the Investigator.
7. Vital signs or clinically significant laboratory values at the screening visit that in the opinion of the Investigator would make the subject an inappropriate candidate for the study.
8. Has taken any other investigational drug during the 30 days prior to the screening visit or is currently participating in another investigational clinical trial.
9. Made any significant donation (including plasma) or have had a significant loss of blood within 30 or 90 days prior to Period 1, Day 1.
10. History or manifestation of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematologic or other medical disorders.
11. Subjects who are carriers of the Hepatitis B surface antigen (HbsAg), Hepatitis C antibody, or HIV antibody.
12. Serious mental or physical illness within the past year.
13. Male subjects who consume more than 28 units of alcohol per week and female subjects who consume more than 21 units of alcohol per week (one unit of alcohol equals 250 mL of beer, 100 mL or a medium glass of wine, or 25 mL of spirits) or those subjects who have a significant history of alcoholism or drug/ chemical abuse within the last 2 years.
14. Failure to agree to abstain from alcohol, cola, tea, coffee, chocolate and other caffeinated drink/ food from 2 days before each dosing and throughout confinement.
15. Positive results on screening tests for drugs of abuse, cotinine or alcohol at screening or the pre-dose assessment at check-in.
16. Subjects who have used tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within 12 months prior to Period 1, Day 1.
17. Women of childbearing potential who are pregnant (as based on test results) or are breast feeding.
18. Subjects who have a history of hypersensitivity or idiosyncratic reaction to any of the products administered during the study.
19. Subjects who, in the opinion of the Investigator, should not participate in the study.
20. Subjects who have a history of unexplained syncope; i.e., autonomic dysfunction.
21. Subjects who have a history of hypotension, including orthostatic hypotension.
22. Lack of ability to understand verbal and/ or written Norwegian.
23. History of severe hypersensitivity or allergic reaction to study medication.
24. Failure to agree to abstain from grapefruit and grapefruit juice as well as oranges and orange juice from 10 days before the first dose and throughout the study.
25. History of clinically significant illness within 4 weeks prior to Day 1.
26. Receipt of a transfusion or any blood products within 90 days prior to Period 1, Day 1.
27. History of participation in another investigational study or who have participated in an investigational study within the past 30 days prior to Period 1, Day 1.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 24 hours after dosing
  To assess the Number of Participants with Adverse Events after dosing, as a Measure of Safety and Tolerability
Pharmacokinetic | 24 hours after dosing
  To assess the pharmacokinetic profiles of theophylline and bambuterol when administered alone or in combination.
  PK sample collections for plasma Theophylline and Bambuterol determinations at 0-hour (pre-dose), and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Trond-Eirik Strand, M.D., Ph.D., Principal Investigator — Institute of Aviation Medicine, Norwegian Armed Forces Medical; Thies Schroeder, Ph.D., Study Director — Department of Radiation Oncology, Duke University Medical Center
Locations (1):
- Institute of Aviation Medicine, Norwegian Armed Forces Medica, Oslo, Norway